CLINICAL TRIAL: NCT05842395
Title: The Role of Vitamin c Supplementation in the Prevention of CRPS Following Distal Radius Fractures: a Randomized Control Study
Brief Title: Vitamin c Supplementation in the Prevention of CRPS Following Distal Radius Fractures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UDMS-Orthopedics-5-2023
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Distal Radius Fracture; Vitamine c; Prophylaxis
Keywords: distal radius fractures; vitamine c; prophylaxis
MeSH Terms: conditions — Wrist Fractures | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants and the consultants making definite treatment decisions and the researcher assistant collecting participants' data will be unaware of allocation until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with distal radius fractures taking vitamin c supplementation. (Experimental): Participants who give informed consent and successfully pass the eligibility criteria will take 1g of oral vitamin C daily for three months.
  Interventions: Drug: Vitamin C
- Participants with distal radius fractures taking a placebo. (Placebo Comparator): Participants who give informed consent and successfully pass the eligibility criteria will take a placebo daily for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — Participants with distal radius fractures will take vitamin C supplementation with a daily dose of 1g orally for three months.
  Arms: Participants with distal radius fractures taking vitamin c supplementation.
Drug: Placebo — Participants with distal radius fractures will take daily Placebo orally for three months.
  Arms: Participants with distal radius fractures taking a placebo.

SUMMARY:
Complex Regional Pain Syndrome type 1 is a pain syndrome that develops after a trauma, surgery, or idiopathically. The incidence after distal radius varies significantly in the literature. There are known contributing factors, such as the female sex but no effective treatment or prophylactic method. This study aims to investigate vitamin C's efficacy in preventing CRPS type 1 following distal radius fractures, as the literature states that it might play a role in prophylaxis.

DETAILED DESCRIPTION:
Complex regional pain syndrome is the most challenging complication to overcome following distal radius fractures. The precise etiology still needs to be fully understood. It is thought that ways of prevention could be the most effective way of managing this dilemma, as no effective treatment is yet to be found.

One of the ways of prevention is vitamin C supplementation, as it is thought that the toxic oxygen radicals play a significant role in the inflammatory process that ultimately manifests as CRPS. Vitamin C, as an antioxidant, could play a role in stopping this process.

The theoretical background of this research is that CRPS commonly occurs following distal radius fractures, and vitamin C supplementation could play a role in prophylaxis. To assess that, the investigator is conducting a randomized controlled trial.

The trial is designed as a multicenter, randomized, controlled study. Two hospitals in Syria, Damascus, participated in this study using the same experimental design.

Adults (18 years or above) with distal radius fractures who will be seen in the emergency department of each hospital will be asked to participate in this study. Patients will be asked to start the trial medication on the day of the fracture following the suitable treatment method chosen by the orthopedics consultant in each hospital. Capsules had to be taken once daily for 90 days. Patients will be allocated randomly to receive either a placebo or 1g of vitamin C daily.

The study's endpoint will be defined as the presence of CRPS at any moment up to one year after the fracture. All participants and physicians will be unaware of the treatment allocation.

The diagnosis will be built upon the Budapest criteria, which will be checked in every follow-up for one year.

Patients will be seen after two weeks, four weeks (or when the cast was removed), six weeks, 12 weeks, six months, and 12 months. The protocol will not compromise the adequate fracture treatment, either conservative or operative, by closed reduction and percutaneous pinning. If necessary, patients will be seen more often and at other times than planned.

ELIGIBILITY:
Inclusion Criteria:

* participants who were injured with distal radius fractures and classified using the AO classification as A1, A2, A3, B1, and C1.

Exclusion Criteria:

* Multiple trauma patients.
* patients who have neurovascular injuries.
* Patients with fractures are classified using the AO classification as B2, B3, C2, and C3.
* Patients who are eligible for open reduction internal fixation of their fractures.
* Patients with chronic or acute renal failure.
* Patients who already take multi-vitamin supplementation or vitamin C supplementation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked 2 weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked four weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked six weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked eight weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked twelve weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked sixteen weeks after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked six months after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.
The positivity of BUDAPEST CRITERIA for diagnosis of CRPS. | checked twelve months after definitive treatment.
  BUDAPEST CRITERIA will be checked for the diagnosis of CRPS type 1.

CONTACTS AND LOCATIONS:
Overall Officials: jaber ibrahim, MD PHD, Study Chair — Damascus university - faculty of medicine - department of surgery; hakam alasaad, MD, Study Director — Damascus university - faculty of medicine - department of surgery; doried Diri, MD, Principal Investigator — Damascus university - faculty of medicine - department of surgery
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pogue DJ, Viegas SF, Patterson RM, Peterson PD, Jenkins DK, Sweo TD, Hokanson JA. Effects of distal radius fracture malunion on wrist joint mechanics. J Hand Surg Am. 1990 Sep;15(5):721-7. doi: 10.1016/0363-5023(90)90143-f. PMID 2229966
- [Background] Sandroni P, Benrud-Larson LM, McClelland RL, Low PA. Complex regional pain syndrome type I: incidence and prevalence in Olmsted county, a population-based study. Pain. 2003 May;103(1-2):199-207. doi: 10.1016/s0304-3959(03)00065-4. PMID 12749974
- [Background] Beerthuizen A, Stronks DL, Van't Spijker A, Yaksh A, Hanraets BM, Klein J, Huygen FJPM. Demographic and medical parameters in the development of complex regional pain syndrome type 1 (CRPS1): prospective study on 596 patients with a fracture. Pain. 2012 Jun;153(6):1187-1192. doi: 10.1016/j.pain.2012.01.026. Epub 2012 Mar 3. PMID 22386473
- [Background] Besse JL, Gadeyne S, Galand-Desme S, Lerat JL, Moyen B. Effect of vitamin C on prevention of complex regional pain syndrome type I in foot and ankle surgery. Foot Ankle Surg. 2009;15(4):179-82. doi: 10.1016/j.fas.2009.02.002. Epub 2009 Apr 5. PMID 19840748
- [Background] van der Laan L, Kapitein PJ, Oyen WJ, Verhofstad AA, Hendriks T, Goris RJ. A novel animal model to evaluate oxygen derived free radical damage in soft tissue. Free Radic Res. 1997 Apr;26(4):363-72. doi: 10.3109/10715769709097816. PMID 9167941
- [Background] Cummings SR, Kelsey JL, Nevitt MC, O'Dowd KJ. Epidemiology of osteoporosis and osteoporotic fractures. Epidemiol Rev. 1985;7:178-208. doi: 10.1093/oxfordjournals.epirev.a036281. No abstract available. PMID 3902494
- [Background] Owen RA, Melton LJ 3rd, Johnson KA, Ilstrup DM, Riggs BL. Incidence of Colles' fracture in a North American community. Am J Public Health. 1982 Jun;72(6):605-7. doi: 10.2105/ajph.72.6.605. PMID 7072880
- [Background] Colles A. On the Fracture of the Carpal Extremity of the Radius. Edinb Med Surg J. 1814 Apr 1;10(38):182-186. No abstract available. PMID 30329360
- [Background] Ilyas AM, Jupiter JB. Distal radius fractures--classification of treatment and indications for surgery. Orthop Clin North Am. 2007 Apr;38(2):167-73, v. doi: 10.1016/j.ocl.2007.01.002. PMID 17560399
- [Background] Muller ME, Nazarian S, Koch PP. Classification AO des fractures. springer; 1987.
- [Background] McKay SD, MacDermid JC, Roth JH, Richards RS. Assessment of complications of distal radius fractures and development of a complication checklist. J Hand Surg Am. 2001 Sep;26(5):916-22. doi: 10.1053/jhsu.2001.26662. PMID 11561246
- [Background] Bushnell BD, Bynum DK. Malunion of the distal radius. J Am Acad Orthop Surg. 2007 Jan;15(1):27-40. doi: 10.5435/00124635-200701000-00004. PMID 17213380
- [Background] Mathews AL, Chung KC. Management of complications of distal radius fractures. Hand Clin. 2015 May;31(2):205-15. doi: 10.1016/j.hcl.2014.12.002. Epub 2015 Feb 28. PMID 25934197
- [Background] Zyluk A, Puchalski P. Complex regional pain syndrome of the upper limb: a review. Neurol Neurochir Pol. 2014;48(3):200-5. doi: 10.1016/j.pjnns.2014.05.007. Epub 2014 Jun 6. PMID 24981185
- [Background] Goris RJ, Dongen LM, Winters HA. Are toxic oxygen radicals involved in the pathogenesis of reflex sympathetic dystrophy? Free Radic Res Commun. 1987;3(1-5):13-8. doi: 10.3109/10715768709069764. PMID 3508426
- [Background] Oaklander AL, Rissmiller JG, Gelman LB, Zheng L, Chang Y, Gott R. Evidence of focal small-fiber axonal degeneration in complex regional pain syndrome-I (reflex sympathetic dystrophy). Pain. 2006 Feb;120(3):235-243. doi: 10.1016/j.pain.2005.09.036. Epub 2006 Jan 19. PMID 16427737
- [Background] Bruehl S, Harden RN, Galer BS, Saltz S, Backonja M, Stanton-Hicks M. Complex regional pain syndrome: are there distinct subtypes and sequential stages of the syndrome? Pain. 2002 Jan;95(1-2):119-24. doi: 10.1016/s0304-3959(01)00387-6. PMID 11790474
- [Background] Zyluk A. [Chronic, refractory algodystrophy]. Chir Narzadow Ruchu Ortop Pol. 2006;71(6):439-46. Polish. PMID 17585487
- [Background] Puchalski P, Zyluk A. Complex regional pain syndrome type 1 after fractures of the distal radius: a prospective study of the role of psychological factors. J Hand Surg Br. 2005 Dec;30(6):574-80. doi: 10.1016/j.jhsb.2005.06.023. Epub 2005 Aug 29. PMID 16126313
- [Background] Perez MRSG, Zuurmond AWW, Bezemer DP, Kuik JD, van Loenen CA, de Lange JJ, Zuidhof JA. The treatment of complex regional pain syndrome type I with free radical scavengers: a randomized controlled study. Pain. 2003 Apr;102(3):297-307. doi: 10.1016/S0304-3959(02)00414-1. PMID 12670672
- [Background] Zyluk A, Puchalski P. Treatment of early complex regional pain syndrome type 1 by a combination of mannitol and dexamethasone. J Hand Surg Eur Vol. 2008 Apr;33(2):130-6. doi: 10.1177/1753193408087034. PMID 18443050
- [Background] Zollinger PE, Tuinebreijer WE, Kreis RW, Breederveld RS. Effect of vitamin C on frequency of reflex sympathetic dystrophy in wrist fractures: a randomised trial. Lancet. 1999 Dec 11;354(9195):2025-8. doi: 10.1016/S0140-6736(99)03059-7. PMID 10636366
- [Background] Abdullah M, Jamil RT, Attia FN. Vitamin C (Ascorbic Acid). 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK499877/ PMID 29763052